CLINICAL TRIAL: NCT05495100
Title: A Single-arm, Multicenter, Prospective Clinical Study of Mitoxantrone Hydrochloride Liposome Injection Combined With Chidamide and Azacitidine in the Treatment of Relapsed and Refractory Peripheral T-cell Lymphoma
Brief Title: A Single-arm, Multicenter, Prospective Clinical Study of Mitoxantrone Liposome Combined With Chidamide and Azacitidine in the Treatment of Relapsed and Refractory Peripheral T-cell Lymphoma
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Collaborators: Ningbo No. 1 Hospital (Other); Jinhua Central Hospital (Other); Huizhou Municipal Central Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2022-0453
Record Dates: First submitted 2022-08-09; First posted 2022-08-10 (Actual); Last update posted 2022-08-10 (Actual); Status verified 2022-08

CONDITIONS: Peripheral T Cell Lymphoma
Keywords: Relapsed and refractory peripheral T-cell lymphoma; mitoxantrone liposomes
MeSH Terms: conditions — Lymphoma, T-Cell, Peripheral; Recurrence

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Mitoxantrone liposome combined with Chidamide and Azacitidine (Experimental)
  Interventions: Drug: Mitoxantrone liposome、Chidamide、Azacitidine

INTERVENTIONS:
Drug: Mitoxantrone liposome、Chidamide、Azacitidine — Mitoxantrone liposome 20mg/m2, d1; Chidamide 20mg, biw; Azacitidine 100mg, d1~7; Every 4 weeks is a cycle, with a maximum of 4 cycles of treatment.

SUMMARY:
To evaluate the efficacy and safety of mitoxantrone hydrochloride liposome injection combined with chidamide and azacitidine in the treatment of relapsed and refractory peripheral T-cell lymphoma

ELIGIBILITY:
Inclusion Criteria:

1. Patients fully understand this study, voluntarily participate in and sign an informed consent form (ICF);
2. Age: 18~75 years old;
3. Expected survival time ≥ 3 months;
4. Histopathologically confirmed PTCL, one of the following subtypes:

(1) Peripheral T-cell lymphoma unspecified (PTCL-NOS) (2) Angioimmunoblastic T-cell lymphoma (AITL) (3) Anaplastic large T-cell lymphoma (ALCL), ALK+ (4) Anaplastic large T-cell lymphoma (ALCL), ALK- (5) Other subtypes of PTCL that the researchers believe can be enrolled; 5. Relapsed/refractory patients who have received at least first-line systemic therapy with anthracycline-containing regimens in the past. Relapse was defined as relapse after CR or progression after PR; refractory was defined as previous systemic chemotherapy treatment, 2 cycles of response evaluation as PD, or 4 cycles of response evaluation as SD; 6. There must be at least one evaluable or measurable lesion that meets the Lugano2014 criteria: lymph node lesions, measurable lymph nodes should be >1.5cm in length; non-lymph node lesions, measurable extranodal lesions should be >1.0cm in length; 7. ECOG score 0-2 points; 8. Bone marrow function: neutrophil count ≥1.5×109/L, platelet count ≥75×109/L, hemoglobin ≥80g/L (the neutrophil count in patients with bone marrow involvement can be relaxed to ≥1.0×109/L, Platelet count can be relaxed to ≥50×109/L, and hemoglobin can be relaxed to ≥75 g/L); Liver and kidney function: Serum creatinine ≤1.5 times the upper limit of normal; AST and ALT ≤2.5 times the upper limit of normal (for patients with liver involvement ≤5 times the upper limit of normal); total bilirubin ≤1.5 times the upper limit of normal (for liver involvement patients ≤ 3 times the upper limit of normal);

Exclusion Criteria:

1. The subject's previous history of anti-tumor therapy meets one of the following conditions:

   1. Those who have received mitoxantrone or mitoxantrone liposome in the past;
   2. Have received doxorubicin or other anthracycline therapy in the past, and the total cumulative dose of doxorubicin is more than 360 mg/m2 (1 mg doxorubicin equivalent to 2 mg epirubicin converted from other anthracyclines);
   3. Patients who have received autologous hematopoietic stem cell transplantation within 100 days of the first medication, or have received allogeneic hematopoietic stem cell transplantation;
   4. Received anti-tumor therapy (including chemotherapy, targeted therapy, hormone therapy, taking traditional Chinese medicine with anti-tumor activity, etc.) or participated in other clinical trials and received clinical trial drugs within 4 weeks before the first use of the study drug;
2. Hypersensitivity to any study drug or its components;
3. Uncontrollable systemic diseases (such as advanced infection, uncontrollable hypertension, diabetes, etc.);
4. Cardiac function and disease meet one of the following conditions:

   1. Long QTc syndrome or QTc interval >480 ms;
   2. Complete left bundle branch block, second or third degree atrioventricular block;
   3. severe, uncontrolled arrhythmia requiring medical treatment;
   4. New York College of Cardiology classification ≥ grade III;
   5. Cardiac ejection fraction (LVEF) less than 50%;
   6. History of myocardial infarction, unstable angina, severe unstable ventricular arrhythmia, or any other arrhythmia requiring treatment, clinically significant pericardial disease within 6 months prior to recruitment, or acute ischemic or active ECG evidence of conduction system abnormalities.
5. Active infection of hepatitis B and C (HBV surface antigen positive and hepatitis B virus DNA more than 1x103 copies/mL; hepatitis C virus RNA more than 1x103 copies/mL);
6. Human immunodeficiency virus (HIV) infection (HIV antibody positive);
7. Past or present with other malignant tumors (except for effectively controlled non-melanoma skin basal cell carcinoma, breast/cervical carcinoma in situ, and other malignant tumors that have been effectively controlled without treatment within the past five years);
8. Suffering from primary or secondary central nervous system (CNS) lymphoma or a history of CNS lymphoma at the time of recruitment;
9. There are obvious gastrointestinal diseases at the time of screening, which may affect the intake, transport or absorption of drugs (such as inability to swallow, chronic diarrhea, intestinal obstruction, etc.);
10. Pregnant, lactating women and patients of childbearing age who are unwilling to take contraceptive measures;
11. Subjects with lymphoma and leukemia (proportion of malignant tumor cells in bone marrow examination> 20%) Circumstances judged by other investigators to be inappropriate to participate in this study. -

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2022-08-11 (Estimated); Primary Completion 2023-08-11 (Estimated); Study Completion 2024-08-11 (Estimated)

PRIMARY OUTCOMES:
ORR | one year
  objective response rate

CONTACTS AND LOCATIONS:
Overall Officials: Wenbin Qian, Principal Investigator — 13605801032
Locations (1):
- Second Affiliated Hospital, School of Medicine, Zhejiang University, Zhejiang, Zhejiang, China